CLINICAL TRIAL: NCT02321397
Title: Randomised, Double-blind, Double-dummy, Cross-over Multicenter Study to Demonstrate Equivalence in Analgesic Efficacy & Bowel Function Taking Oxycodone Equivalents of 120 & 160 mg Per Day as Achieved With the Higher OXN PR Tablet Strengths (OXN60/30 mg PR, OXN80/40 mg PR) BID Compared to the Identical Daily Dose Taken as a Combination of Lower Tablet Strengths in Subjects With Non-malignant or Malignant Pain That Requires Around-the-clock Opioid Therapy.
Brief Title: To Demonstrate Equivalence in Analgesic Efficacy & Bowel Function Between OXN PR Higher Dose & Lower Dose Tablet Strengths in Subjects With Non-cancer or Cancer Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OXN3508; 2013-004888-31 (EudraCT Number)
Record Dates: First submitted 2014-10-13; First posted 2014-12-22 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2015-12

CONDITIONS: Malignant Pain; Non-malignant Pain
Keywords: oxycodone naloxone combination; severe chronic and non-malignant pain; Malignant and non-malignant pain that requires around-the clock opioid therapy
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OXN PR HST (Experimental): Prolonged release oxycodone/naloxone higher strength tablets
  Interventions: Drug: Oxycodone
- OXN PR LST (Active Comparator): Prolonged release oxycodone/naloxone lower strength tablets
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Oxycodone
  Arms: OXN PR HST
Drug: Naloxone — Prolonged Release Tablets
  Arms: OXN PR LST

SUMMARY:
This study is aimed to demonstrate equivalence between combinations of lower strength OXN PR tablets (OXN PR LST) and single higher strength OXN PR tablets (OXN PR HST) taken at the same overall daily dose.

DETAILED DESCRIPTION:
Study OXN3508 is a multicenter double-blind, double-dummy, randomised, cross-over, 2-period, phase III study in male and female subjects with severe non-malignant or malignant pain that requires around-the-clock opioid therapy at a daily dose of 120/60 mg or 160/80 mg oxycodone/naloxone prolonged release (OXN PR).

ELIGIBILITY:
Inclusion Criteria

* Subjects who are receiving WHO step III opioid analgesic medication for the treatment of non-malignant or malignant pain.
* Documented history of non-malignant or malignant pain that requires around-the-clock opioid therapy

Exclusion Criteria

* Females who are pregnant or lactating.
* Subjects with evidence or significant structural abnormalities of the gastrointestinal tract.
* Subjects with evidence of impaired liver/kidney function upon entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
(mean of subjects average pain over the last 24 hours as assessed by the pain intensity scale.) | 24 hours at one day in week 2, 3 5 and 6 from date of randomisation.
  Pain scores based on the mean of subjects average pain over the last 24 hours as assessed by the pain intensity scale. To demonstrate equivalence between multiple lower strength OXN PR tablets and a single higher strength OXN PR tablet taken at the same overall total daily dose
Equivalent bowel function as assessed by the Bowel Function Index (BFI). | Week 2, 3 5 and 6 from date of randomisation.

SECONDARY OUTCOMES:
Pain scores of subjects average pain over the last 24 hours and rescue medication use. | Week 1,2,3,4,5 and 6 from date of randomisation
To assess bowel function (assess BFI and laxative use) | Week 1,2,3,4,5 and 6 from date of randomisation
  To assess BFI and laxative use
To assess quality of life based on the EuroQol EQ-5D. | Visit 3 and visit 6 from date of randomisation
  EuroQol EQ-5D is a standardized instrument for use as a measure of health outcome.
Number of participants with adverse events, high/low laboratory values and clinically significant ECG findings. | Up to 35 weeks
Pain right now scores at intake of oxycodone/naloxone tablets. | Week 2,3,5 and 6 from date of randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- Mainz, Germany